CLINICAL TRIAL: NCT06988891
Title: Effects of 'Evidence-based Practice' Training Based on Flipped Learning, Web-based and Traditional Education Models on Nurses' Self-directed Learning and Metacognitive Thinking Skills
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Deniz Yilidirim, MSc, BSN, PhD Student in the Department of Education in Nursing, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IstanbulUC-RN-02; Istanbul University Cerrahpasa (Other: Istanbul University Cerrahpasa)
Record Dates: First submitted 2025-05-12; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Flipped Education Model; Self Directed Learning; Metacognition; Web Based Education
Keywords: nursing education; self directed learning; metacognition; flipped learning

STUDY DESIGN:
Intervention Model Description: A randomised controlled experimental study with a pre-test-post-test design consisting of two intervention groups (flipped learning and web-based training) and one control group (traditional training).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Evidence-based practice training based on the flipped learning model (Experimental): Evidence-based practice training developed based on the flipped learning model was applied to the nurses in this group once a week for four weeks.
  Interventions: Other: 'Evidence-based practice' training based on the flipped learning model
- 'Evidence-based practice' training based on web-based education model (Active Comparator): Evidence-based practice training developed based on the WEB-based education model was applied to the nurses in this group once a week for two weeks.
  Interventions: Other: 'Evidence-based practice' training based on web-based education model
- 'Evidence-based practice' training based on traditional education model (Placebo Comparator): Evidence-based practice training, developed based on the traditional/face-to-face education model, was applied to the nurses in this group once a week for three weeks.
  Interventions: Other: 'Evidence-based practice' training based on traditional education model

INTERVENTIONS:
Other: 'Evidence-based practice' training based on the flipped learning model — The evidence-based practice training, developed using the flipped learning model, was delivered once a week for four weeks. Each session was delivered as an offline training (3-24 February 2025) and a face-to-face training three days later (6-27 February 2025). The offline part of the training was delivered via the Edpuzzle platform. The training duration for each session was 75 minutes in total, 15 minutes offline and 60 minutes face-to-face.
  Arms: Evidence-based practice training based on the flipped learning model
Other: 'Evidence-based practice' training based on web-based education model — Evidence-based practice training, developed based on a web-based training model, was implemented once a week for two weeks (March 17-24, 2025). Each session was conducted offline. The first session was 20.10 minutes, and the second session was 17.44 minutes.
  Arms: 'Evidence-based practice' training based on web-based education model
Other: 'Evidence-based practice' training based on traditional education model — The evidence-based practice training, developed based on the traditional/face-to-face education model, was delivered once a week for three weeks (7-21 April 2025). Each session consisted of two teaching hours (one teaching hour: 45 minutes).
  Arms: 'Evidence-based practice' training based on traditional education model

SUMMARY:
The research was conducted to evaluate the effects of evidence-based practice training developed based on flipped learning, web-based education and traditional education models on nurses' self-directed learning and metacognitive thinking skills. The study is a randomised controlled experimental study with a pre-test-post-test design, consisting of two intervention groups (flipped learning and web-based education) and one control group (traditional education).

DETAILED DESCRIPTION:
Purpose: The purpose of the study is to evaluate the effects of evidence-based practice training developed based on flipped learning, web-based education and traditional education models on nurses' self-directed learning and metacognitive thinking skills.

Method: The study is a pre-test-post-test randomised controlled experimental research design with two intervention groups (flipped learning and web-based education models applied) and one control group (traditional education model applied). The study was conducted with 45 nurses working in a training and research hospital in Istanbul. Data were collected with self-directed learning skills and metacognitive thinking skills scales.

ELIGIBILITY:
Inclusion Criteria:

* Have at least a bachelor's degree in nursing

Exclusion Criteria:

* Requesting to withdraw from the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Self Directed Learning Skills Scale | one month
  The scale was developed to determine the self-directed learning skill levels of learners. It consists of 21 items and 4 sub-dimensions (self-monitoring, motivation, self-control, self-confidence). The response options of the five-point Likert-type scale are; "(1) Never to (5) Always." The highest score that can be obtained from the scale is 105, the middle score is 63, and the lowest score is 21. An increase in the score obtained from the scale indicates that the participant has high self-directed learning skills. The total Cronbach α value of the scale was determined as 0.91 in the study.

SECONDARY OUTCOMES:
Metacognitive thinking skills scale | one month
  It was developed to determine the metacognitive thinking skills levels of individuals. The scale consists of 18 items and 4 sub-dimensions (thinking skills, reflective thinking skills for problem solving, decision-making skills, alternative assessment skills). The response options of the five-point Likert-type scale are from (1) Totally disagree to (5) Totally agree. The highest score that can be obtained from the scale is 90, the lowest score is 18. An increase in the score obtained from the scale indicates that metacognitive thinking skills have increased. The total Cronbach α value of the scale was determined as 0.90 in the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Taşcıoğlu Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biyik Bayram S, Gulnar E, Ozveren H, Caliskan N. The effect of flipped learning on blood pressure knowledge and self-directed learning skills of first-year nursing students: A randomized controlled trial. Nurse Educ Pract. 2023 Feb;67:103557. doi: 10.1016/j.nepr.2023.103557. Epub 2023 Jan 25. PMID 36709659